CLINICAL TRIAL: NCT00926432
Title: 3D Evaluation of Postural Balance of the Adult Affected by Postural Trouble, Using EOS™ Images and 3D-reconstructions With Regard to Gravity Line.
Brief Title: Postural Balance of the Adult
Acronym: POSTURADULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: EOS imaging Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2008/32
Record Dates: First submitted 2009-06-18; First posted 2009-06-23 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Postural Balance
Keywords: Balance; Spine disorders; equilibrium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Other): Small group of aged healthy volunteers
  Interventions: Device: EOS™ Acquisition
- Patients (Other): Patients consulting for spine disorders that may or may not have postural troubles
  Interventions: Device: EOS™ Acquisition

INTERVENTIONS:
Device: EOS™ Acquisition — Double Incidence Postero Anterior and Lateral full body low-dose X-ray acquisition on EOS™ device following SOP of the service of radiology.
  Arms: Healthy volunteers
Device: EOS™ Acquisition — Double Incidence Postero Anterior and Lateral full body low-dose X-ray acquisition on EOS™ device following SOP of the service of radiology.
  Arms: Patients

SUMMARY:
Description of the geometrical configuration of the skeleton with regard to gravity line by patients suffering from spinal disorders that may induce postural troubles

DETAILED DESCRIPTION:
In clinical routine, 3D analysis of postural balance is only made using clinical examination. When dealing with specific pathologies, in particular spine disorders, a better understanding of the balance could help better treat and prevent late complications. This prospective study aims at describing the pathologies of the musculoskeletal system using 3D reconstruction of the spine, the pelvis and the inferior limbs with regard to gravity line by patients suffering from postural trouble and defining new parameters to assess postural balance

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to social insurance
* Informed of the benefits, the risks and the conduction of the study and have given their free informed consent.

For Patients

* Medical prescription for an EOS™ exam, or for Frontal AND Lateral full-spine radiographs or for a pangonogram.

For Healthy Volunteers

* 50 years old

Exclusion Criteria:

For Patients

* Patients that neither need any EOS™ exam, nor Face & Lateral full-spine radiographs, nor pangonogram.

For Healthy Volunteers

* Children or young adults (<50)
* Psychiatric or neurologic deficit.
* Anterior Surgery of Spine or inferior Member
* Chronic back pain
* Recent acute back Pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the three-dimensional geometrical configuration of the skeleton with respect to the gravity line on a large population of patient presenting a broad spectrum of pathologies inducing postural imbalance. | 1 day

SECONDARY OUTCOMES:
3D Position of the middle of acoustic meati, of each vertebral body, of the center of both acetabula and the barycentre of the four condyles with respect to the gravity line. | 1 day
Morphologic and positioning parameters of the pelvis (pelvic incidence, pelvic version, sacral slope & pelvic radius) | 1 day
Kyphosis, lordosis and sinopelvic balance | 1 day
To validate the measure of femoral and tibial torsion using EOS™ images | 1 day
influence of position change on the evaluation of changes in postural balance following surgery | After surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc VITAL, Professor, Principal Investigator — Hospital University, Bordeaux; Wafa SKALLI, PhD, Pr, Study Director — Laboratoire de Biomécanique Arts et Metiers ParisTech-CNRS UMR 8005
Locations (1):
- Unité de Pathologie Rachidienne Tripode CHU Pellegrin, Place Amélie Raba-Léon, Bordeaux, France

REFERENCES:
- [Background] Dubousset J, Charpak G, Skalli W, Kalifa G, Lazennec JY. [EOS stereo-radiography system: whole-body simultaneous anteroposterior and lateral radiographs with very low radiation dose]. Rev Chir Orthop Reparatrice Appar Mot. 2007 Oct;93(6 Suppl):141-3. doi: 10.1016/s0035-1040(07)92729-4. No abstract available. French. PMID 18033112
- [Background] Schwab F, Lafage V, Boyce R, Skalli W, Farcy JP. Gravity line analysis in adult volunteers: age-related correlation with spinal parameters, pelvic parameters, and foot position. Spine (Phila Pa 1976). 2006 Dec 1;31(25):E959-67. doi: 10.1097/01.brs.0000248126.96737.0f. PMID 17139212
- [Background] Skalli W, Zeller RD, Miladi L, Bourcereau G, Savidan M, Lavaste F, Dubousset J. Importance of pelvic compensation in posture and motion after posterior spinal fusion using CD instrumentation for idiopathic scoliosis. Spine (Phila Pa 1976). 2006 May 20;31(12):E359-66. doi: 10.1097/01.brs.0000219402.01636.87. PMID 16721280
- [Background] El Fegoun AB, Schwab F, Gamez L, Champain N, Skalli W, Farcy JP. Center of gravity and radiographic posture analysis: a preliminary review of adult volunteers and adult patients affected by scoliosis. Spine (Phila Pa 1976). 2005 Jul 1;30(13):1535-40. doi: 10.1097/01.brs.0000167534.49069.e9. PMID 15990669
- [Background] Rillardon L, Campana S, Mitton D, Skalli W, Feydy A. [Evaluation of the intervertebral disc spaces with a low dose radiographic system]. J Radiol. 2005 Mar;86(3):311-9. doi: 10.1016/s0221-0363(05)81360-5. French. PMID 15908871
- [Background] Dubousset J, Charpak G, Dorion I, Skalli W, Lavaste F, Deguise J, Kalifa G, Ferey S. [A new 2D and 3D imaging approach to musculoskeletal physiology and pathology with low-dose radiation and the standing position: the EOS system]. Bull Acad Natl Med. 2005 Feb;189(2):287-97; discussion 297-300. French. PMID 16114859
- [Background] Vialle R, Levassor N, Rillardon L, Templier A, Skalli W, Guigui P. Radiographic analysis of the sagittal alignment and balance of the spine in asymptomatic subjects. J Bone Joint Surg Am. 2005 Feb;87(2):260-7. doi: 10.2106/JBJS.D.02043. PMID 15687145
- [Background] Parent S, Labelle H, Skalli W, de Guise J. Vertebral wedging characteristic changes in scoliotic spines. Spine (Phila Pa 1976). 2004 Oct 15;29(20):E455-62. doi: 10.1097/01.brs.0000142430.65463.3a. PMID 15480123
- [Background] Faro FD, Marks MC, Pawelek J, Newton PO. Evaluation of a functional position for lateral radiograph acquisition in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2004 Oct 15;29(20):2284-9. doi: 10.1097/01.brs.0000142224.46796.a7. PMID 15480143
- [Background] Steib JP, Dumas R, Mitton D, Skalli W. Surgical correction of scoliosis by in situ contouring: a detorsion analysis. Spine (Phila Pa 1976). 2004 Jan 15;29(2):193-9. doi: 10.1097/01.BRS.0000107233.99835.A4. PMID 14722414
- [Background] Gangnet N, Pomero V, Dumas R, Skalli W, Vital JM. Variability of the spine and pelvis location with respect to the gravity line: a three-dimensional stereoradiographic study using a force platform. Surg Radiol Anat. 2003 Nov-Dec;25(5-6):424-33. doi: 10.1007/s00276-003-0154-6. Epub 2003 Sep 16. PMID 13680185
- [Background] Dumas R, Steib JP, Mitton D, Lavaste F, Skalli W. Three-dimensional quantitative segmental analysis of scoliosis corrected by the in situ contouring technique. Spine (Phila Pa 1976). 2003 Jun 1;28(11):1158-62. doi: 10.1097/01.BRS.0000068242.29809.D0. PMID 12782985
- [Background] Rajnics P, Templier A, Skalli W, Lavaste F, Illes T. The association of sagittal spinal and pelvic parameters in asymptomatic persons and patients with isthmic spondylolisthesis. J Spinal Disord Tech. 2002 Feb;15(1):24-30. doi: 10.1097/00024720-200202000-00004. PMID 11891447
- [Background] Legaye J, Duval-Beaupere G, Hecquet J, Marty C. Pelvic incidence: a fundamental pelvic parameter for three-dimensional regulation of spinal sagittal curves. Eur Spine J. 1998;7(2):99-103. doi: 10.1007/s005860050038. PMID 9629932
- [Background] Jackson RP, Peterson MD, McManus AC, Hales C. Compensatory spinopelvic balance over the hip axis and better reliability in measuring lordosis to the pelvic radius on standing lateral radiographs of adult volunteers and patients. Spine (Phila Pa 1976). 1998 Aug 15;23(16):1750-67. doi: 10.1097/00007632-199808150-00008. PMID 9728376
- [Background] Gelb DE, Lenke LG, Bridwell KH, Blanke K, McEnery KW. An analysis of sagittal spinal alignment in 100 asymptomatic middle and older aged volunteers. Spine (Phila Pa 1976). 1995 Jun 15;20(12):1351-8. PMID 7676332
- [Background] Mitton D, Zhao K, Bertrand S, Zhao C, Laporte S, Yang C, An KN, Skalli W. 3D reconstruction of the ribs from lateral and frontal X-rays in comparison to 3D CT-scan reconstruction. J Biomech. 2008;41(3):706-10. doi: 10.1016/j.jbiomech.2007.09.034. Epub 2007 Nov 5. PMID 17981286
- [Background] Rousseau MA, Laporte S, Chavary-Bernier E, Lazennec JY, Skalli W. Reproducibility of measuring the shape and three-dimensional position of cervical vertebrae in upright position using the EOS stereoradiography system. Spine (Phila Pa 1976). 2007 Nov 1;32(23):2569-72. doi: 10.1097/BRS.0b013e318158cba2. PMID 17978655
- [Background] Gille O, Champain N, Benchikh-El-Fegoun A, Vital JM, Skalli W. Reliability of 3D reconstruction of the spine of mild scoliotic patients. Spine (Phila Pa 1976). 2007 Mar 1;32(5):568-73. doi: 10.1097/01.brs.0000256866.25747.b3. PMID 17334292
- [Background] Hemophilia: state of the art in 1982. Vox Sang. 1983;45(1):93-5. doi: 10.1159/000466070. No abstract available. PMID 6880151
- [Background] Dumas R, Aissaoui R, Mitton D, Skalli W, de Guise JA. Personalized body segment parameters from biplanar low-dose radiography. IEEE Trans Biomed Eng. 2005 Oct;52(10):1756-63. doi: 10.1109/TBME.2005.855711. PMID 16235661
- [Background] Le Bras A, Laporte S, Bousson V, Mitton D, De Guise JA, Laredo JD, Skalli W. 3D reconstruction of the proximal femur with low-dose digital stereoradiography. Comput Aided Surg. 2004;9(3):51-7. doi: 10.3109/10929080400018122. PMID 15792937
- [Background] Pomero V, Mitton D, Laporte S, de Guise JA, Skalli W. Fast accurate stereoradiographic 3D-reconstruction of the spine using a combined geometric and statistic model. Clin Biomech (Bristol). 2004 Mar;19(3):240-7. doi: 10.1016/j.clinbiomech.2003.11.014. PMID 15003338
- [Background] Parent S, Labelle H, Skalli W, de Guise J. Thoracic pedicle morphometry in vertebrae from scoliotic spines. Spine (Phila Pa 1976). 2004 Feb 1;29(3):239-48. doi: 10.1097/01.brs.0000109995.64028.fe. PMID 14752344
- [Background] Dumas R, Le Bras A, Champain N, Savidan M, Mitton D, Kalifa G, Steib JP, de Guise JA, Skalli W. Validation of the relative 3D orientation of vertebrae reconstructed by bi-planar radiography. Med Eng Phys. 2004 Jun;26(5):415-22. doi: 10.1016/j.medengphy.2004.02.004. PMID 15147749
- [Background] Le Bras A, Laporte S, Mitton D, de Guise JA, Skalli W. 3D detailed reconstruction of vertebrae with low dose digital stereoradiography. Stud Health Technol Inform. 2002;91:286-90. PMID 15457739
- [Background] Laporte S, Skalli W, de Guise JA, Lavaste F, Mitton D. A biplanar reconstruction method based on 2D and 3D contours: application to the distal femur. Comput Methods Biomech Biomed Engin. 2003 Feb;6(1):1-6. doi: 10.1080/1025584031000065956. PMID 12623432
- [Background] Mitulescu A, Skalli W, Mitton D, De Guise JA. Three-dimensional surface rendering reconstruction of scoliotic vertebrae using a non stereo-corresponding points technique. Eur Spine J. 2002 Aug;11(4):344-52. doi: 10.1007/s00586-002-0432-8. Epub 2002 Jun 26. PMID 12193996
- [Background] Mitulescu A, Semaan I, De Guise JA, Leborgne P, Adamsbaum C, Skalli W. Validation of the non-stereo corresponding points stereoradiographic 3D reconstruction technique. Med Biol Eng Comput. 2001 Mar;39(2):152-8. doi: 10.1007/BF02344797. PMID 11361240
- [Background] Kalifa G, Charpak Y, Maccia C, Fery-Lemonnier E, Bloch J, Boussard JM, Attal M, Dubousset J, Adamsbaum C. Evaluation of a new low-dose digital x-ray device: first dosimetric and clinical results in children. Pediatr Radiol. 1998 Jul;28(7):557-61. doi: 10.1007/s002470050413. PMID 9662585